CLINICAL TRIAL: NCT02996682
Title: A Multicenter, Randomized, Phase 3, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir ± Ribavirin for 12 Weeks in Subjects With Chronic HCV Infection and Decompensated Cirrhosis
Brief Title: Efficacy and Safety of Sofosbuvir/Velpatasvir ± Ribavirin for 12 Weeks in Adults With Chronic HCV Infection and Decompensated Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-4019
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Virus Infection
Keywords: Communicable Diseases; Hepatitis; Hepatitis C; Virus Diseases; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Velpatasvir; RNA Virus Infections; Ribavirin; Sofosbuvir; Antiviral Agents; Antimetabolites; Molecular Mechanisms of Pharmacological Action; Anti-Infective Agents; Decompensated Cirrhosis
MeSH Terms: conditions — Hepatitis C; Communicable Diseases; Hepatitis; Virus Diseases; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; RNA Virus Infections | interventions — sofosbuvir-velpatasvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOF/VEL (Experimental): SOF/VEL for 12 weeks
  Interventions: Drug: SOF/VEL
- SOF/VEL + RBV (Experimental): SOF/VEL + RBV for 12 weeks
  Interventions: Drug: SOF/VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®
Drug: RBV — Capsules administered orally in a divided daily dose
  Other Names: Rebetol®
  Arms: SOF/VEL + RBV

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) with or without ribavirin (RBV) for 12 weeks in adults with chronic hepatitis C virus (HCV) infection and decompensated cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV-infected males and non-pregnant/non-lactating females
* Treatment naive or treatment experienced individuals
* Child-Pugh-Turcotte Score 7-12 at screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-12-26 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (33):
- Japan (33):
  - Shimonoseki, Yamaguchi
  - Bunkyō City
  - Chiba
  - Chūō
  - Ehime
  - Fukui
  - Fukuyama-shi
  - Hiroshima
  - Ibaraki
  - Ichikawa
  - Iizuka
  - Iruma
  - Izunokuni
  - Kashibara
  - Kofu
  - Kumamoto
  - Kurume
  - Kyoto
  - Miyazaki
  - Morioka
  - Musashino
  - Nagoya
  - Nishinomiya
  - Okayama
  - Osaka
  - Ōmura
  - Sapporo
  - Sendai
  - Shimotsuga-gun
  - Suita
  - Takamatsu
  - Ube
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Result] Takehara T, Kurosaki M, Tanaka Y, Tatsumi T, Ikeda F, Takikawa Y, et al. Sofosbuvir/Velpatasvir with or without Ribavirin for 12 Weeks in HCV-Infected Japanese Subjects with Decompensated Cirrhosis [Presentation]. 54th Annual Meeting of Japan Society of Hepatology; 2018 June 15; Osaka, Japan.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 26 December 2016. The last study visit occurred on 08 May 2018.
Pre-assignment Details: 155 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks
- SOF/VEL + RBV: SOF/VEL (400/100 mg) FDC tablet once daily + ribavirin (RBV) capsules (600, 800, or 1,000 mg daily based on weight and CPT class) for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL | SOF/VEL + RBV
Started | 51 | 51
Completed | 51 | 48
Not Completed | 0 | 3
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet once daily for 12 weeks
- SOF/VEL + RBV: SOF/VEL (400/100 mg) FDC tablet once daily + RBV capsules (600, 800, or 1,000 mg daily based on weight and CPT class) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL | SOF/VEL + RBV | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66 (9.6) | 66 (9.6) | 66 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 29 | 62
  Male | 18 | 22 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 51 | 51 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1 | 41 | 39 | 80
  Genotype 2 | 9 | 11 | 20
  Genotype 3 | 1 | 0 | 1
  Missing | 0 | 1 | 1
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 33 | 37 | 70
    CT | 16 | 13 | 29
    TT | 2 | 1 | 3
HCV RNA (log10 international units per milliliter [IU/mL]) [Mean (Standard Deviation); unit: log10 IU/mL] | 5.7 (0.70) | 5.8 (0.55) | 5.8 (0.63)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 30 | 30 | 60
  ≥ 800,000 IU/mL | 21 | 21 | 42
Model for End Stage Liver Disease (MELD) Score Category [Count of Participants; unit: Participants] — MELD score is a chronic liver disease severity scoring system. Scores can range from 6 to 40, with higher scores indicating greater disease severity.
  Participants
    < 10 MELD Score | 10 | 15 | 25
    10-15 MELD Score | 36 | 33 | 69
    16-20 MELD Score | 4 | 2 | 6
    21-25 MELD Score | 0 | 1 | 1
    > 25 MELD Score | 1 | 0 | 1
Child-Pugh-Turcotte (CPT) Class [Count of Participants; unit: Participants] — CPT is a chronic liver disease classification system. Classes include CPT Class A, CPT Class B, and CPT Class C, in order of greater disease severity. During screening/randomization, CPT scores may have been assessed using either the international normalized ratio (INR) or prothrombin activation percentage for the coagulation parameter.
  Participants
    CPT A [5-6] | 1 | 2 | 3
    CPT B [7-9] | 40 | 39 | 79
    CPT C [10-15] | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants | 92.2 [81.1 to 97.8] | 92.2 [81.1 to 97.8]
Statistical Analysis 1: Comparison: SOF/VEL; A sample size of 50 participants in each treatment group would provide over 99% power to detect at least 40% improvement in SVR12 rate from the assumed spontaneous rate of 1% or less using a 2-sided exact 1-sample binomial test at significance level of 0.025; Test type: Superiority; p < 0.001, 2-sided exact 1-sample binomial test — P-value was from the 2-sided exact 1-sample binomial test for the superiority of each treatment group over pre-specified rate of 1%
Statistical Analysis 2: Comparison: SOF/VEL + RBV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, 2-sided exact 1-sample binomial test — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Participants Who Discontinued Treatment (SOF/VEL or RBV) Early Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants
  Discontinuation of SOF/VEL | 0 | 3.9
  Discontinuation of RBV | NA — RBV drug was not used an as intervention in this arm. | 17.6

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants | 94.1 [83.8 to 98.8] | 96.1 [86.5 to 99.5]

4. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants | 92.2 [81.1 to 97.8] | 92.2 [81.1 to 97.8]

5. Secondary Outcome: Percentage of Participants Who Had HCV RNA < LLOQ by Visit While on Treatment
Time Frame: Up to 12 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants
  Week 2 | 45.1 | 51.0
  Week 4 | 96.1 | 90.2
  Week 8 | 100.0 | 96.1
  Week 12: number analyzed (Participants) | 51 | 49
  Week 12 | 100.0 | 100.0

6. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline and up to 12 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
log10 IU/mL
  Change at Week 2 | -4.14 (0.573) | -4.33 (0.525)
  Change at Week 4 | -4.55 (0.696) | -4.65 (0.528)
  Change at Week 8: number analyzed (Participants) | 51 | 49
  Change at Week 8 | -4.56 (0.705) | -4.70 (0.554)
  Change at Week 12: number analyzed (Participants) | 51 | 49
  Change at Week 12 | -4.56 (0.705) | -4.70 (0.554)

7. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase in Model for End Stage Liver Disease (MELD) Score
Description: MELD score is a chronic liver disease severity scoring system. Scores can range from 6 to 40, with higher scores indicating greater disease severity. "No change" was assigned for differences (posttreatment visits minus baseline score) of -1, 0 or 1; "Decrease" was assigned for differences that were less than or equal to -2; and "Increase" was assigned for values that were greater than or equal to 2.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set who achieved SVR24 with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 47 | 46
Percentage of participants
  Decrease (Improvement) | 38.3 | 21.7
  No Change | 53.2 | 54.3
  Increase (Worsening) | 8.5 | 23.9

8. Secondary Outcome: Percentage of Participants With Improved and Worsened Child-Pugh-Turcotte (CPT) Class
Description: CPT is a chronic liver disease classification system. Classes include CPT Class A, CPT Class B, and CPT Class C, in order of greater disease severity. Participants with improved CPT class was defined as having Class C at Baseline and Class B or A at Posttreatment Week 24 or Class B at Baseline and Class A at Posttreatment Week 24. Participants with worsened CPT class was defined as having Class A at Baseline and Class B or C at Posttreatment Week 24 or Class B at Baseline and Class C at Posttreatment Week 24. CPT scores were calculated using prothrombin activation percentage for the coagulation parameter per Japan's standard.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set who achieved SVR24 with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 47 | 46
Percentage of participants
  Improved CPT Class | 36.2 | 39.1
  Worsened CPT Class | 4.3 | 2.2

9. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment), or Relapse (HCV RNA ≥ LLOQ during the post-treatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available post-treatment measurement).
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL | SOF/VEL + RBV
Number analyzed (Participants) | 51 | 51
Percentage of participants | 7.8 | 3.9

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 12 weeks plus 30 days; All-Cause Mortality: Up to Posttreatment Week 24
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | SOF/VEL | SOF/VEL + RBV
All-Cause Mortality (participants affected / at risk) | 0/51 | 3/51
Serious Adverse Events (participants affected / at risk) | 4/51 | 7/51
Other Adverse Events (participants affected / at risk) | 14/51 | 34/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=51) | SOF/VEL + RBV (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=51) | SOF/VEL + RBV (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 19
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 7
Oedema peripheral (General disorders) | 3 | 2
Nasopharyngitis (Infections and infestations) | 7 | 3
Gastroenteritis (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Headache (Nervous system disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02996682/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/82/NCT02996682/SAP_001.pdf